CLINICAL TRIAL: NCT04539184
Title: The Effectiveness and Cost-effectiveness of Motion Style Acupuncture Treatment (MSAT) for Acute Neck Pain: A Multi-center Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2020-08
Record Dates: First submitted 2020-08-26; First posted 2020-09-04 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Acute Neck Pain
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motion Style Acupuncture treatment (Experimental): Motion Style Acupuncture treatment (2-3 times/week, 2 weeks)
  Interventions: Other: Motion Style Acupuncture Treatment (MSAT)
- Acupuncture treatment (Active Comparator): Acupuncture treatment (2-3 times/week, 2 weeks)
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Motion Style Acupuncture Treatment (MSAT) — MSAT required a part of the patient's body to move passively or actively while acupuncture needles are retained.
  Arms: Motion Style Acupuncture treatment
Other: Acupuncture — General acupuncture
  Arms: Acupuncture treatment

SUMMARY:
The investigators will evaluate the comparative effectiveness and safety of Motion Style Acupuncture Treatment (MSAT) therapy for acute neck pain compared to acupuncture.

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled, comparative effectiveness clinical trial for acute neck pain. Motion style acupuncture requires a part of the patient's body to move passively or actively while acupuncture needles are retained.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain onset or worsen within one month
* VAS of neck pain on movement or at rest of 5 or higher
* Age between 19 and 70 years old
* Participants who wrote a informed consent

Exclusion Criteria:

* Participants who diagnosed with the serious disease that can cause pain (e.g. Migration of cancer reaching to spine, fracture of spine, dislocation of spine)
* Progressive neurologic deficits or severe neurologic deficits
* Participants who diagnosed with a soft tissue disease that can cause pain (Cancer, fibromyalgia, RA, or goat)
* Chronic disease (e.g. Cardiovascular disease, kidney disease, dementia, diabetic neuropathy, or epilepsy)
* Participants taking steroids, immunosuppressants, or psychotropic medication
* Participants who could be inadequate or unsafe at acupuncture (e.g. Hemorrhagic disease, severe diabetes or taking anticoagulant drug)
* Participants who took NSAIDs or acupuncture within 3 days
* Participants who had undergone cervical surgery within 3 months
* Participants who had a traffic accident within a month
* Pregnant or women who planned to conceive
* Participants who had participated in other clinical trial within 1 month, or have plan for participation in other trial within 6 months from enrollment
* Participants who can not write informed consent
* Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale(VAS) on movement | Change from baseline VAS at 3 weeks
  Minimum 0, Maximum 100. Higher values represent a worse outcome

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) on movement | Baseline(Week 1), Week 2, 3, 8
  Minimum 0, Maximum 100. Higher values represent a worse outcome
Visual Analogue Scale (VAS) at rest | Baseline(Week 1), Week 2, 3, 8
  Minimum 0, Maximum 100. Higher values represent a worse outcome
Numeric Rating Scale (NRS) on movement | Baseline(Week 1), Week 2, 3, 8
  Minimum 0, Maximum 10. Higher values represent a worse outcome
Numeric Rating Scale (NRS) at rest | Baseline(Week 1), Week 2, 3, 8
  Minimum 0, Maximum 10. Higher values represent a worse outcome
Vernon-Mior Neck Disability Index (NDI) | Baseline(Week 1), Week 2, 3, 8
  Functional disability questionnaire
Northwick Park Neck Pain Questionnaire (NPQ) | Baseline(Week 1), Week 2, 3, 8
  Functional disability questionnaire and Pain questionnaire
Patient Global Impression of Change (PGIC) | Week 3, 8
  Global, patient-reported outcome, Minimum 1, Maximum 7, Higher values represent a better outcome
Range of movement (ROM) of flexion | Baseline(Week 1), Week 2, 3, 8
  Range of movement of flexion
Range of movement (ROM) of extension | Baseline(Week 1), Week 2, 3, 8
  Range of movement of extension
Range of movement (ROM) of Rt rotation | Baseline(Week 1), Week 2, 3, 8
  Range of movement of Right rotation
Range of movement (ROM) of Lt rotation | Baseline(Week 1), Week 2, 3, 8
  Range of movement of Left rotation
Range of movement (ROM) of Lt lateroflexion | Baseline(Week 1), Week 2, 3, 8
  Range of movement of Left lateroflexion
Range of movement (ROM) of Rt lateroflexion | Baseline(Week 1), Week 2, 3, 8
  Range of movement of Right lateroflexion
EQ-5D-5L | Baseline(Week 1), 3, 8
  Health-related quality of life questionnaire
12-item Short-Form Health Survey (SF-12) | Baseline(Week 1), 3, 8
  Health-related quality of life questionnaire
EuroQol Visual Analogue Scale (EQ-VAS) | Baseline(Week 1), 3, 8
  Health-related quality of life questionnaire
Adverse events | Time Frame: Baseline (Week 1), Week 2, 3, 8 (every visit)
  Safety outcome
Drug Consumption | Time Frame: Baseline (Week 1), Week 2, 3, 8 (every visit)
  Drug type and dose of prescribe for medicine or rescue medicine, and type and frequency of other treatments

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Dr., Principal Investigator — Jaseng Medical Foundation
Locations (4):
- South Korea (4):
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YJ, Kim D, Park KS, Kim S, Seo JY, Cho HW, Heo I, Shin WC, Cho JH, Kim JH, Seo BK, Ha IH. Effectiveness and safety of motion style acupuncture treatment for acute neck pain: a multicenter randomized controlled trial. Chin Med. 2026 Jan 23;21(1):49. doi: 10.1186/s13020-026-01332-0. PMID 41572363
- [Derived] Kim D, Lee YJ, Park KS, Kim S, Seo JY, Cho HW, Ha IH. The effectiveness and cost-effectiveness of motion style acupuncture treatment (MSAT) for acute neck pain: A multi-center randomized controlled trial. Medicine (Baltimore). 2020 Oct 30;99(44):e22871. doi: 10.1097/MD.0000000000022871. PMID 33126334